CLINICAL TRIAL: NCT02053129
Title: Pilot Evaluation of Pulmonary Tuberculosis Screening in Antenatal Clinics in Lusaka, Zambia
Brief Title: Evaluation of PTB Screening in ANC in Lusaka, Zambia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Centre for Infectious Disease Research in Zambia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CIDRZ 1217/IRB12-0417
Record Dates: First submitted 2014-01-31; First posted 2014-02-03 (Estimated); Last update posted 2017-09-15 (Actual); Status verified 2014-12

CONDITIONS: Pulmonary Tuberculosis
Keywords: tuberculosis; HIV; pregnancy
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis | interventions — Culture Techniques; Single Person

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HIV negative pregnant women (Other): Pregnant women who are HIV negative attending their first ANC visit
  Interventions: Other: TB screening Questionnaire
- HIV positive pregnant women (Other): Pregnant women who are HIV positive accessing antenatal care.
  Interventions: Other: TB screening Questionnaire; Other: Sputum smear and culture (only in HIV negative women who are symptomatic)

INTERVENTIONS:
Other: TB screening Questionnaire — All subjects will be screened with the questionnaire which assesses TB symptoms.
  Other Names: Pilot TB symptom questionnaire
Other: Sputum smear and culture (only in HIV negative women who are symptomatic) — specimens for sputum microscopy and culture collected and processed in accordance with WHO TB Infection Control Guidelines
  Arms: HIV positive pregnant women

SUMMARY:
This is a pilot pulmonary TB screening program done in three antenatal care clinics in Lusaka, Zambia to determine the prevalence of culture-confirmed pulmonary tuberculosis and to determine the sensitivity and specificity of symptom-based TB screening.

DETAILED DESCRIPTION:
5000 pregnant women attending antenatal clinics will be evaluated by piloting a TB symptom questionnaire as part of the general health screening done at each visit. Due to the atypical and subclinical presentation of TB in HIV infected patients, culture will be performed on all HIV-infected pregnant women, with or without symptoms, and on all symptomatic HIVnegative women. Referrals for TB treatment in accordance with current national guidelines will be offered.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* 18 years or older
* HIV-negative women with any TB symptoms or HIV-infected women regardless of TB symptoms
* Attending first ANC visit at one of program clinics

Exclusion Criteria:

* HIV negative without any TB symptoms

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5033 (Actual)
Dates: Start 2011-11; Primary Completion 2012-10 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
number of positive pulmonary tuberculosis (PTB) tests | 1 day of screening (first antenatal visit)
  The prevalence of culture confirmed PTB among HIV positive and HIV negative pregnant women will be measured to determine if there is a substantial amount of undiagnosed TB in the HIV positive population accessing antenatal care.

SECONDARY OUTCOMES:
Sensitivity and specificity of symptom-based TB screening | 1 day of screening visit
  To determine the sensitivity and specificity of symptom based TB screening (compared to TB culture), enrollees will have TB symptoms assessed by administration of a questionnaire. Culture will then be performed on all HIV infected pregnant women, with or without symptoms, and on all symptomatic HIV negative women.

CONTACTS AND LOCATIONS:
Overall Officials: Stewart Reid, MD, Principal Investigator — Centre for Infectious Disease Research in Zambia; Nzali Kancheya, MMED, MPH, Principal Investigator — Centre for Infectious Disease Research in Zambia; Michael Saag, MD, Principal Investigator — Professor, University of Alabama; German Henostroza, MD, Principal Investigator — Centre for Infectious Disease Research in Zambia; Annika Kruuner, MD, Principal Investigator — Centre for Infectious Disease Research in Zambia
Locations (1):
- Centre for Infectious Disease Research in Zambia, Lusaka, Zambia

REFERENCES:
- [Background] Global tuberculosis control: Epidemiology, Strategy, Financing. WHO report 2009. 2009, World Health Organization: Geneva, Switzerland.
- [Background] Black V, Brooke S, Chersich MF. Effect of human immunodeficiency virus treatment on maternal mortality at a tertiary center in South Africa: a 5-year audit. Obstet Gynecol. 2009 Aug;114(2 Pt 1):292-299. doi: 10.1097/AOG.0b013e3181af33e6. PMID 19622990
- [Background] Mwaba P, Maboshe M, Chintu C, Squire B, Nyirenda S, Sunkutu R, Zumla A. The relentless spread of tuberculosis in Zambia--trends over the past 37 years (1964-2000). S Afr Med J. 2003 Feb;93(2):149-52. PMID 12640889
- [Background] WHO. TB Country Profile for Zambia: Surveillance and Epidemiology. 2009 [cited; Available from: http://apps.who.int/globalatlas/predefinedReports/TB/PDF_Files/zmb.pdf
- [Background] Ayles H, Schaap A, Nota A, Sismanidis C, Tembwe R, De Haas P, Muyoyeta M, Beyers N; Peter Godfrey-Faussett for the ZAMSTAR Study Team. Prevalence of tuberculosis, HIV and respiratory symptoms in two Zambian communities: implications for tuberculosis control in the era of HIV. PLoS One. 2009;4(5):e5602. doi: 10.1371/journal.pone.0005602. Epub 2009 May 19. PMID 19440346
- [Background] Tripathy SN, Tripathy SN. Tuberculosis and pregnancy. Int J Gynaecol Obstet. 2003 Mar;80(3):247-53. doi: 10.1016/s0020-7292(02)00393-4. PMID 12628525
- [Background] Murray CJ, Lopez AD. Mortality by cause for eight regions of the world: Global Burden of Disease Study. Lancet. 1997 May 3;349(9061):1269-76. doi: 10.1016/S0140-6736(96)07493-4. PMID 9142060
- [Background] Harries AD, Parry C, Nyongonya Mbewe L, Graham SM, Daley HM, Maher D, Salaniponi FM, Nyangulu DS. The pattern of tuberculosis in Queen Elizabeth Central Hospital, Blantyre, Malawi: 1986-1995. Int J Tuberc Lung Dis. 1997 Aug;1(4):346-51. PMID 9432391
- [Background] Khan M, Pillay T, Moodley JM, Connolly CA; Durban Perinatal TB HIV-1 Study Group. Maternal mortality associated with tuberculosis-HIV-1 co-infection in Durban, South Africa. AIDS. 2001 Sep 28;15(14):1857-63. doi: 10.1097/00002030-200109280-00016. PMID 11579249
- [Background] WHO. Fact Sheet- Women and TB; 2009. 2009 [cited; Available from: http://www.stoptb.org/resource_center/assets/factsheets/womenandtb.pdf
- [Background] Pillay T, Khan M, Moodley J, Adhikari M, Padayatchi N, Naicker V, Pillay DG, Coovadia HM. The increasing burden of tuberculosis in pregnant women, newborns and infants under 6 months of age in Durban, KwaZulu-Natal. S Afr Med J. 2001 Nov;91(11):983-7. PMID 11847922
- [Background] Celine R. Gounder, M., ScM*, Nikolas Wada, MPH*, Caroline Kensler, MHS*, Avy Violari, MD**, Richard E. Chaisson, MD*, James McIntyre, MBChB, FRCOG***, Neil Martinson, MBChB, MPH*,**, Provider-Initiated Screening for Tuberculosis (TB) among Pregnant Women in Antenatal Clinics in Soweto, South Africa, in 17th Conference on Retroviruses and Opportunistic Infections. 2010: San Francisco, CA. February 16 - 19 2010.
- [Background] Kali PB, Gray GE, Violari A, Chaisson RE, McIntyre JA, Martinson NA. Combining PMTCT with active case finding for tuberculosis. J Acquir Immune Defic Syndr. 2006 Jul;42(3):379-81. doi: 10.1097/01.qai.0000218434.20404.9c. PMID 16645548
- [Background] Gupta A, Nayak U, Ram M, Bhosale R, Patil S, Basavraj A, Kakrani A, Philip S, Desai D, Sastry J, Bollinger RC; Byramjee Jeejeebhoy Medical College-Johns Hopkins University Study Group. Postpartum tuberculosis incidence and mortality among HIV-infected women and their infants in Pune, India, 2002-2005. Clin Infect Dis. 2007 Jul 15;45(2):241-9. doi: 10.1086/518974. Epub 2007 Jun 4. PMID 17578786
- [Background] Ahmed Y, Mwaba P, Chintu C, Grange JM, Ustianowski A, Zumla A. A study of maternal mortality at the University Teaching Hospital, Lusaka, Zambia: the emergence of tuberculosis as a major non-obstetric cause of maternal death. Int J Tuberc Lung Dis. 1999 Aug;3(8):675-80. PMID 10460099
- [Background] Margono F, Mroueh J, Garely A, White D, Duerr A, Minkoff HL. Resurgence of active tuberculosis among pregnant women. Obstet Gynecol. 1994 Jun;83(6):911-4. doi: 10.1097/00006250-199406000-00001. PMID 8190429
- [Background] Bjerkedal T, Bahna SL, Lehmann EH. Course and outcome of pregnancy in women with pulmonary tuberculosis. Scand J Respir Dis. 1975;56(5):245-50. PMID 1209197
- [Background] Figueroa-Damian R, Arredondo-Garcia JL. Pregnancy and tuberculosis: influence of treatment on perinatal outcome. Am J Perinatol. 1998 May;15(5):303-6. doi: 10.1055/s-2007-993948. PMID 9643636
- [Background] Jana N, Vasishta K, Jindal SK, Khunnu B, Ghosh K. Perinatal outcome in pregnancies complicated by pulmonary tuberculosis. Int J Gynaecol Obstet. 1994 Feb;44(2):119-24. doi: 10.1016/0020-7292(94)90064-7. PMID 7911094
- [Background] Pillay T, Khan M, Moodley J, Adhikari M, Coovadia H. Perinatal tuberculosis and HIV-1: considerations for resource-limited settings. Lancet Infect Dis. 2004 Mar;4(3):155-65. doi: 10.1016/S1473-3099(04)00939-9. PMID 14998501
- [Background] Amita Gupta, N.G., Sandesh Patil, Pradeep Sambarey, Sandhya Khadse, Anju Kagal, Suvarna Joshi, Arun Jamkar, Robert Bollinger, and the SWEN India Study Group1Johns, Maternal TB is associated with increased risk of HIV mother-to-child transmission, in 17th Conference on Retroviruses and Opportunistic Infections. 2010: San Francisco, CA. February 16 - 19 2010
- See also: University of North Carolina website — http://www.unc.edu